CLINICAL TRIAL: NCT01895920
Title: Viral Biofilms: Hijacking T Cell Extracellular Matrix to Regulate HIV-1 Spread?
Acronym: TRANSBioHIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ANRS RF001 TRANSBioHIV
Record Dates: First submitted 2013-07-02; First posted 2013-07-11 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2017-05

CONDITIONS: HIV Infection
Keywords: HIV; Biofilm; Transmission
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV infection (Experimental): 20 HIV infected subjects
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample

SUMMARY:
This project aims at characterizing HIV-1 viral biofilms structural and functional properties and at deciphering its role as a new viral reservoir and as a new mode of viral spread. The prospective national study will be conducted on cells isolated from blood samples from 20 patients infected with HIV.

DETAILED DESCRIPTION:
The investigators' preliminary data indicate that besides " free " infectious viral particles, HIV-1 infected cluster of differentiation 4 (CD4+) lymphocytes also produce extracellular viral assemblies wrapped in an extracellular matrix cocoon and tightly bound to the surface of the cell. Importantly, these structures are infectious, transferred to target cells upon intercellular contacts and they are key role in HIV-1 spread between T lymphocytes. HIV-1 viral biofilm could be important not only for direct transmission of the virions but also for " trans-infection ", a process our objectives are:

* to better characterize the molecular composition and the architecture of this biofilm (using proteomics, glycomic superresolution cell imaging approaches) with regard to its properties (infectivity, adhesiveness, protection of virions) and to determine whether cells from infected patients produce such structures.
* to delineate the viral factors regulating the formation of these new infectious structures (with a particular attention on Tat, Vpu and Nef HIV-1 encoded using mutant viruses or expression vectors).
* to investigate the lymphocyte pathways regulating the viral biofilms formation and composition in extracellular matrix (ECM) proteins (using quantitative polymerase chain reaction (qPCR) and siRNA).
* to determine whether those viral biofilms are involved in HIV-1 transmission by transinfection
* to study the contribution of those infectious structures and the dynamics of their transmission in lymph nodes.

This project may contribute to decipher the role of viral biofilms in HIV-1 transmission. Ultimately, we intend to determine how the interference of retroviral infections with T cell activation pathways modulates the pattern of ECM production by T cells, tuning viral biofilm composition and regulating viral dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* able to give written consent
* HIV positive serology HIV1
* Viral load > 10 000 copies/ml
* CD4 T cells > 100 cells/mm3
* or Treated by antiretroviral therapy (ARV) for less than 6 months
* Covered by French Social Security

Exclusion Criteria:

* Involved in a clinical trial
* Pregnancy (inclusion can be postponed)
* No covered by French Social Security

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The percentage of HIV positive patients with cells producing biofilms. | 2 years

SECONDARY OUTCOMES:
The number of cells with biofilms identified among the HIV positive patients presenting such structures. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Interne, CHU Kremlin-Bicêtre, Le Kremlin-Bicêtre, France